CLINICAL TRIAL: NCT02705989
Title: A Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics(PK) and Pharmacodynamics(PD), and Non-Randomized, Bioavailability(BA) Study of BMS-986195 in Healthy Subjects
Brief Title: Safety, Tolerability and Relative Bioavailability Study of BMS-986195 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM014-001
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — branebrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single Ascending Dose (SAD) (Placebo Comparator): Single ascending dose of BMS-986195 or Placebo matching BMS-986195
  Interventions: Drug: BMS-986195; Other: Placebo
- Multiple Ascending Dose(MAD) (Placebo Comparator): Multiple ascending dose of BMS-986195 or Placebo matching BMS-986195
  Interventions: Drug: BMS-986195; Other: Placebo
- Japanese-Multiple Ascending Dose(MAD) (Placebo Comparator): Multiple ascending dose of BMS-986195 or Placebo matching BMS-986195 in subjects with Japanese heritage
  Interventions: Drug: BMS-986195; Other: Placebo
- Relative Bioavailability with Food Effects (Open Label) (Experimental)
  Interventions: Drug: BMS-986195

INTERVENTIONS:
Drug: BMS-986195 — Specified dose on specified day
Other: Placebo — Specified dose on specified day
  Arms: Japanese-Multiple Ascending Dose(MAD); Multiple Ascending Dose(MAD); Single Ascending Dose (SAD)

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, pharmacokinetics, and pharmacodynamics following single and multiple ascending oral doses of BMS-986195 in healthy subjects, and to assess the relative bioavailability of two formulations of BMS-986195 with or without food.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body Mass Index(BMI) of 18 to 32 kilograms/meter^2
* Healthy male and female, first generation Japanese with confirmed paternal and maternal Japanese ancestry, 18-55 years old, whose residency outside of Japan does not exceed 10 years with a BMI of 18-30 kilograms/meter^2 inclusive.
* Women must not be pregnant or breastfeeding
* Women of Childbearing Potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 14 days or longer if required.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 14 days or longer if required.

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Known or suspected autoimmune disorder, including but not limited to rheumatoid arthritis, fibromyalgia, systemic lupus erythematosis, polymyalgia rheumatica, giant cell arteritis, Behcet's disease, dermatomyositis, multiple sclerosis, moderate to severe asthma, any autoimmune vasculitis, autoimmune hepatitis, or any other active autoimmune disease for which a subject requires medical follow-up or medical treatment
* Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the subject's immune status (example: history of splenectomy)
* Presence of any factors that would predispose the subject to develop infection e.g., rectal fissures, poor dentition, open skin lesions, and presence of preexisting skin conditions that increase risks for injection site complications e.g. Behcet's Disease, Psoriasis, pustular dermatoses
* Any history or risk for tuberculosis (TB)

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 439 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single oral dose of BMS-986195 as determined by medical review of adverse event reports, vital sign measurements, electrocardiograms (ECGs), and results of physical examination and laboratory tests | Up to 8 days during and after last dose
Safety and tolerability of multiple oral doses of BMS-986195 as determined by medical review of adverse event reports, vital sign measurements, electrocardiograms (ECGs), and results of physical examination and laboratory tests | Up to 21 days during and after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Melbourne, Victoria, Australia

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx